CLINICAL TRIAL: NCT06273956
Title: Assessment of Bleeding Scores in Immune Thrombocytopenia Purpuria
Brief Title: Explore the Relationship Between Platelet Count and Bleeding Score in ITP
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Sayed Hamed, Assistant Lecturer, Assiut University
Other Study IDs: bleeding scores in ItP
Record Dates: First submitted 2024-01-19; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: bleeding scores
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

SUMMARY:
Assessment of bleeding scores in immune thrombocytopenia purpuria to explore the relationship between platelet count and bleeding score in immune thrombocytopenia purpura (ITP) and compare the clinical practicability of bleeding grading systems with adult patients with ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia purpura (ITP) is an autoimmune hemorrhagic disease, characterized by a decreased platelet count ( < 100*109) and suppressed platelet development . The incidence of ITP increases with age, with an incidence rate of 20-40/ million adults (over 18 years old) /year and higher in the people over 60 years old . The main clinical manifestations were bleeding symptoms, but heterogeneity between manifestations was noted. Severe thrombocytopenia is considered as a risk factor for bleeding in ITP, but patients with moderate or even mild thrombocytopenia can also experience severe bleeding, which seems like a disproportionate performance

. Bleeding is one of the leading causes of death in patients with thrombocytopenia . Bleeding manifestations in ITP with mild mucocutaneous to life-threatening bleeding, and prediction of severe bleeding is instructive to the management of thrombocytopenia.

Bleeding assessment tools, such as ITP Bleeding Assessment Tool (ITP-BAT), ITP Bleeding Scale (IBLS) and Khellaf bleeding score, have been developed and studied in a variety of clinical settings for diagnosis and to evaluate the severity of bleeding.

In this study, investigators retrospectively assessed the relationship between platelet count and bleeding score in patients with ITP and compared the clinical aspects of existing ITP bleeding score systems .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary ITP .

Exclusion Criteria:

* Malignancy disease
* Virus infection:

  * HIV
  * Hepatitis B virus
  * Hepatitis C virus
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adults(≥18 years old) , diagnosed as primary ITP
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
explore the relationship between platelet count and bleeding assessment systems (ITP Bleeding Assessment Tool (ITP -BAT) and ITP Bleeding Scale (IBLS) in Patients with ITP to measure severity of bleeding | througth study completion, an average of 3 years
  ITP -BAT :
  Bleeding signs/symptoms are grouped according to three major domains: Skin (S), visible Mucosa (M) and Organs (O).
  Gradation of bleeding severity (SMOG system): Each bleeding manifestation should be assessed at the time of examination. Its severity is graded from 0 to 4. Appreciation of bleeding based on history only, without supporting medical documentation, will be given a grade 1 designation. Within each domain, the same grading is assigned to the symptoms judged to have similar clinical relevance. For each symptom, the worst ever episode during the observation period is graded and then the worst episode within the domain is recorded.
  ITP Bleeding Scale (IBLS) :
  The ITP Bleeding Scale (IBLS) is a novel bleeding assessment system comprising 11 site-specific grades. The IBLS is a useful clinical tool for monitoring bleeding and may be used to aid the development of laboratory parameters that correlate with underlying bleeding propensity in thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Mohammed Mahmoud Hafez, professor, Study Chair — Assiut University; Yousreyia Abdel Rahman Ahmed, professor, Study Chair — Assiut University
Locations (1):
- Aml Sayed Hamed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No